CLINICAL TRIAL: NCT03450070
Title: Repeat Insult Patch Testing (RIPT) APPENDIX I to HRL Standard Protocol #100
Brief Title: Repeat Insult Patch Test APPENDIX I to HRL Standard Protocol #100
Acronym: RIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO- 171028001439-SACT
Record Dates: First submitted 2018-01-19; First posted 2018-03-01 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Allergic Sensitization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Panel (Experimental): Light Therapy Mask Cream
  Interventions: Device: Light Therapy Mask Cream

INTERVENTIONS:
Device: Light Therapy Mask Cream — test panel

SUMMARY:
Patch Testing for device cream on human subjects

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18+ years
* Good health
* Signed and datad Informed Consent
* Signed and dated HIPAA

Exclusion Criteria:

* On test at any other research lab or clinic
* Known allergy or sensitivity to cosmetics or toiletries
* Pre-existing other medical conditions
* Treatment with antibiotics, antihistamines, or corticosteroids within 2 weeks of the test
* Chronic medication which could affect the outcome of the study
* Known pregnant or nursing women
* Cancer diagnosis within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harrison Research Laboratories, Union, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 121 subjects enrolled. 3 of those subjects were disconinued prior to being patched due to screen failure. Therefore, 118 subjects started using patches.
Period: Overall Study
Arm/Group | Test Panel
Started | 118
Completed | 110
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: Only subjects that completed the study per protocol were included in the analysis
Arm/Group | Test Panel
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 105
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Did Not Have Test Material Induced Clinically Significant Dermal Irritation
Description: "Clinically Significant Dermal Irritation" refers to an overall outcome measure in which, after 6 weeks of the test (patching the skin (3 weeks) & then challenging the skin (at week 6)), the test product caused a clinically significant dermal reaction (scores of 2 or greater). Participant scores less than 2 are not considered to be Clinically significant.
  Scoring System:
  0 = No visible reaction
  ± = Faint, minimal erythema
  1. = Erythema
  2. = Intense erythema
  3. = Intense erythema, induration, vesicles
  4. = Severe reaction with erythema, induration, vesicles, pustules (may be weeping) E = Edema DR = Dryness P = Peeling S = Staining
     * = Hyperpigmentation / Hypopigmentation C = Change of test site N9R = No 9th reading
       * = No patch application and / or reading TR = Tape Reaction
Time Frame: approximately 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Test Panel
Number analyzed (Participants) | 110
Participants | 110

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Test Panel
All-Cause Mortality (participants affected / at risk) | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) will provide Sponsor with at least sixty (60) days to review any Publication. No Publication that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, the PI withholds such Publication for up to an additional sixty (60) days to allow for filing of a patent application.

DOCUMENTS (1):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03450070/Prot_000.pdf